CLINICAL TRIAL: NCT03943355
Title: Is Strict Adherence to the Nonoperative Management Protocol Associated With Better Outcome in Patients With Blunt Splenic Injuries
Brief Title: Nonoperative Management Protocol in Patients With Blunt Splenic Injuries
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-4441B
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Blunt Injuries
MeSH Terms: conditions — Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nonoperative management protocol with angioembolization: The nonoperative management (NOM) protocol with angioembolization (AE) presents a trend in dealing with trauma patients with blunt splenic injury (BSI). This study was designed to explore the adverse events and associated risk factors before and after protocol-based NOM of BSI over a 12-year period.
  Interventions: Other: Patient before cohort (2005-2010); Other: Patient after cohort (2011-2016)

INTERVENTIONS:
Other: Patient before cohort (2005-2010) — The NOM protocol with AE was recognized and accepted after our previous study reported in 2004.
Other: Patient after cohort (2011-2016) — The protocol of NOM became more aggressively and strictly adhered to since 2011.

SUMMARY:
This study was designed to explore the adverse events and associated risk factors before and after protocol-based NOM of BSI over a 12-year period in our institution.

DETAILED DESCRIPTION:
The nonoperative management (NOM) protocol with angioembolization (AE) presents a trend in dealing with trauma patients with blunt splenic injury (BSI). This study was designed to explore the adverse events and associated risk factors before and after protocol-based NOM of BSI over a 12-year period.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients with blunt splenic injury who were admitted from 2005 to 2016.

Exclusion Criteria:

* Patients younger than 16 years
* Patients who died in the emergency department

Ages: 17 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective study was performed on adult trauma patients with BSI who were admitted from 2005 to 2016. The patients were divided into before cohort (2005-2010) and after cohort (2011-2016).
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
The numbers of associated complications and mortality | up to 6 months
  The primary outcome of interest in this study would be the associated complications and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: TSANG-TANG Hsieh, MD, Study Chair — Chang Gung Memorial Hospital